CLINICAL TRIAL: NCT06304727
Title: Evaluation of Short Enteral Nutrition and Monitoring in the Emergency Room for Infants Under 1 Year of Age With Bronchiolitis With Main Nutritional Impairment
Brief Title: Evaluation of Short Enteral Nutrition in the Emergency Room for Bronchiolitis With Main Nutritional Impairment
Acronym: 1TreSBCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5064; Easydore (Other: 69HCL23_0736)
Record Dates: First submitted 2024-01-18; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-01

CONDITIONS: Bronchiolitis
Keywords: infant; bronchiolitis; enteral feeding
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- enteral feeding group: Infants < 1 year old with bronchiolitis and exclusive nutritional impairment who underwent short-term enteral feeding and monitoring in the emergency room according to the 2022-2024 seasons protocol
  Interventions: Other: clinical data review

INTERVENTIONS:
Other: clinical data review — Medical records review to gather and analyze demographic, clinical, care and virological data

SUMMARY:
The winter epidemic of bronchiolitis in infants poses insurmountable difficulties for the hospital system for the 2022-2023 season globally. These difficulties are linked to the combination of an unusual epidemic intensity and the loss of medical and paramedical caregivers in the hospital leading to the closure of beds since the Covid-19 pandemic. Bronchiolitis in youngest and most vulnerable infants can lead to severe clinical pictures requiring hospitalization. Among them, some infants present exclusively with inability to eat and only require continuous enteral nutrition during their hospitalization.

A service protocol has been put in place in the pediatric emergency room of the Hôpital Femme Mère Enfant for the 2022-2023 season to carry out short enteral nutrition and monitoring before returning home. This outpatient care would aim to reduce the effect of hospital saturation during the winter epidemic of bronchiolitis, increase the comfort and satisfaction of families by allowing less disruption of family life and prevent nosocomial infections.

A retrospective evaluation of the feasibility and effectiveness of this protocol is necessary to rely on this first experience of outpatient management.

ELIGIBILITY:
Inclusion Criteria:

* Children being treated according to our Short-Term Enteral Nutrition Protocol

Exclusion Criteria:

* Parents refusal

Ages: 8 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Inclusion of all infants under one year old presenting a bronchiolitis with exclusive nutritional impairment and treated in the emergency room of the Hôpital Femme Mère Enfant according to the Protocole de prise en charge de la bronchiolite avec forme digestive prédominante à l'accueil des urgences de l'HFME (Protocol for the management of bronchiolitis with a predominantly digestive form at the HFME emergency department)- ZSBCD. This population will constitute a restrospective cohort in a pediatric tertiary care hospital during the 2022-2023 bronchiolitis season.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the short enteral feeding protocol | From day1 of protocol inclusion
  yes/no Protocol outcome (return home or hospitalization, new short-term consultation)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mere Enfant, Bron, France